CLINICAL TRIAL: NCT06371976
Title: Evaluation of the Hypothalamic-pituitary-adrenal Axis in Patients With Vasoplegic Syndrome After Cardiac Surgery
Brief Title: Evaluation of the HPA Axis in Patients With Vasoplegic Syndrome After Cardiac Surgery
Acronym: VASOCORT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APH240230
Record Dates: First submitted 2024-03-21; First posted 2024-04-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Vasoplegic Syndrome in Adult Cardiac Surgery
Keywords: vasoplegia; vasoplegic shock; cardiac vasoplegia syndrome
MeSH Terms: conditions — Vasoplegia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing cardiac surgery: The patients included will be adult patients scheduled for cardiac surgery with extracorporeal circulation.
  Interventions: Other: Blood sampling; Other: Vital status

INTERVENTIONS:
Other: Blood sampling — Blood samples of 5 mL are taken at 4 stages of the study. Samples are taken from an arterial catheter inserted as part of the treatment, for a total volume of 20 mL maximum for the study.
Other: Vital status — Patients will be followed until their discharge from intensive care, or at most until D28, and their vital status will be collected at the end of their participation in the study.

SUMMARY:
Vasoplegic syndrome after cardiac surgery is common and is associated with increased morbidity and mortality. It is characterized by early and prolonged arterial hypotension, with preserved cardiac output and low systemic vascular resistance. Vasoplegic syndrome therefore shares pathophysiological features with septic shock. There are no data in the literature on the function of the hypothalamic-pituitary-adrenal (HPA) axis during vasoplegic syndrome after cardiac surgery. In situations of acute stress and systemic inflammation, relative adrenal insufficiency has been reported in the most severe patients, particularly those in septic shock. The term ""CIRCI"" (Critical Illness-Related Corticosteroid Insufficiency) is currently defined as an increase in total plasma cortisol of less than 9 µg/dl after stimulation with 250 µg tetracosactide (synthetic ACTH), or a basal total plasma cortisol level of less than 10 µg/dl. However, recent studies have called into question the usefulness of the cosyntropin stimulation test for exploring the HPA axis in intensive care patients.

Tandem mass spectrometry (LC-MS/MS) assays can be used to measure steroid metabolites (steroidome), enabling more precise exploration of the corticotropic axis.

The aim of this study is to evaluate, on an exploratory basis, the impact of the presence of a post-cardiac surgery vasoplegic syndrome on adrenal function by steroidome mapping (LC-MS/MS).

DETAILED DESCRIPTION:
Vasoplegic syndrome after cardiac surgery is common (incidence 5-44%) and is associated with increased morbidity and mortality. It is characterized by early (immediately or within the first 24 hours post-operatively) and prolonged (more than 4 hours) arterial hypotension, with preserved cardiac output and low systemic vascular resistance. Vasoplegic syndrome therefore shares pathophysiological features with septic shock. There are no data in the literature on the function of the hypothalamic-pituitary-adrenal (HPA) during vasoplegic syndrome after cardiac surgery. In situations of acute stress and systemic inflammation, relative adrenal insufficiency has been reported in the most severe patients, particularly those in septic shock. The term ""CIRCI"" (Critical Illness-Related Corticosteroid Insufficiency) is currently defined as an increase in total plasma cortisol of less than 9 µg/dl after stimulation with 250 µg tetracosactide (synthetic ACTH), or a basal total plasma cortisol level of less than 10 µg/dl. However, recent studies have called into question the usefulness of the cosyntropin stimulation test for exploring the HPA axis in intensive care patients. An increase in the volume of cortisol distribution, a decrease in cortisol-binding protein and cortisol clearance (notably via an increase in bile acids) could distort test interpretation: the slight increase in total plasma cortisol would contrast with a normal increase in free cortisol.

Tandem mass spectrometry (LC-MS/MS) assays can be used to measure steroid metabolites (steroidome), enabling more precise exploration of the corticotropic axis. Another study, has shown that steroidome analysis by LC-MS/MS enables the diagnosis of adrenal insufficiency with excellent sensitivity and specificity in a population of women with hyperandrogenism.

The aim of this study is to evaluate, on an exploratory basis, the impact of the presence of a post-cardiac surgery vasoplegic syndrome on adrenal function by steroidome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled cardiac surgery with extracorporeal circulation
* Patient or trusted person or legal representative informed and having expressed non-opposition to participation in the study.

Exclusion Criteria:

* Previous treatment within the last 3 months with glucocorticoids, azoles (Fluconazole, Voriconazole), phenytoin, rifampin, glitazones (Rosiglitazone or Pioglitazone), imipraminics (Clomipramine, Imipramine, Amitriptyline), barbiturates (Primidone, Phenobarbital, Thiopenthal) or phenothiazines (Chlorpromazine, Cyamemazine).
* Adrenal or intracranial pathology affecting the hypothalamic-pituitary axis.
* Cardiac transplants.
* Post-operative mechanical extracorporeal assistance.
* Patient deprived of liberty by judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included will be adult patients scheduled for cardiac surgery with extracorporeal circulation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-02-05 (Estimated)

PRIMARY OUTCOMES:
Impact of post-cardiac surgery vasoplegic syndrome on corticotropic function. | 4 hours post-operatively
  steroidome mapping (LC-MS/MS)

SECONDARY OUTCOMES:
Evaluate corticotropic function by measuring steroid metabolites according to the presence or absence of ""CIRCI"" in patients with vasoplegic syndrome. | between day 0 and day 4
  increase in total plasma cortisol below 9 µg/dl after stimulation with 250 µg IV tetracosactide (synthetic ACTH) or basal total plasma cortisol below 10 µg/dl.
Evaluate the association between CIRCI and the severity of vasoplegic syndrome after cardiac surgery. | up to 28 days
  duration of catecholamine support, maximum vaso-inotropic score in the first 24 hours (VISmaxH24), variation in the Sequential Organ Failure score (ΔH48-SOFA) over the first 48 hours, duration of mechanical ventilation, duration of extra-renal purification, D28 mortality
To assess the association between ""CIRCI"" and the duration of post-cardiac surgery vasoplegic syndrome. | up to 28 days
  Number of days without catecholamines at day 28
To assess the association between ""CIRCI"" and length of stay in intensive care. | up to 28 days
  Length of stay in critical care
Evaluate the association between ""CIRCI"" and in-hospital mortality | up to 28 days
  mortality at day28

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié-Salpêtrière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, "Commission nationale de l'informatique et des libertés") do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.